CLINICAL TRIAL: NCT06237374
Title: Supporting Community Health Workers as Vaccine Educators: Assessing the Impact of a Digital Health Training and Patient-facing Chatbot Intervention on Vaccination Rates in Kenya
Brief Title: Supporting CHWs as Vaccine Educators: Impact of a Digital Training and Chatbot Intervention on Vaccination in Kenya
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jamie Johnston, Research Director, Stanford Center for Health Education, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 69793
Record Dates: First submitted 2024-01-24; First posted 2024-02-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Vaccine Knowledge; Vaccine Hesitancy; Vaccine Refusal
MeSH Terms: conditions — Vaccination Hesitancy; Vaccination Refusal

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized trial with baseline covariate adjustment and stratification. The randomization unit is the Community Health Unit (CHU), the administrative unit in which community health workers (CHWs) are organized in the study region. The randomization will be stratified by geographic unit (wards) and whether a health facility is located in the ward. The following baseline characteristics will be measured and adjusted for in the main analysis of primary outcomes to increase statistical efficiency: 1) age, 2) gender, 3) language, 4) years of work experience, 5) vaccine beliefs, and 6) self-reported preparedness to educate patients about vaccination.
Who Masked: Participant
Masking Description: The CHWs will be blinded to treatment assignment and informed that they are taking part in a study to understand the CHW experiences and their communication with patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Community health workers (CHWs) will receive the intervention training videos, job aids and chatbot tool to share with patients via WhatsApp in addition to standard CHW training provided by Lwala Community Health Alliance.
  Interventions: Behavioral: Digital Vaccine Education Training & Patient-facing Chatbot Tool; Behavioral: Standard Training
- Control (Active Comparator): Participants in the control group will receive standard community health worker (CHW) training provided by Lwala Community Health Alliance.
  Interventions: Behavioral: Standard Training

INTERVENTIONS:
Behavioral: Digital Vaccine Education Training & Patient-facing Chatbot Tool — The first part of the intervention is a digital training provided to CHWs, which includes videos and job aids on vaccine education to support patient communication. The second part of the intervention is a patient-facing chatbot designed to provide key information about routine immunization that CHWs can share with their patients through the social media and messenger application, WhatsApp.
  Arms: Treatment
Behavioral: Standard Training — All CHWs in the study will receive the standard CHW training that is provided on an ongoing basis by Lwala Community Health Alliance.

SUMMARY:
This study seeks to understand how to support community health workers (CHWs) to improve routine vaccination rates in high-need areas by testing a two-part intervention. The first part of the intervention is a digital training provided to CHWs, which includes videos and job aids on vaccine education to support patient communication. The second part of the intervention is a patient-facing chatbot that CHWs can share with their patients. The chatbot is designed to answer patient questions about routine immunization. The intervention will be implemented in two sub-counties in Migori County Kenya (Awendo and Nyatike) that Lwala Community Health Alliance has identified as high need with respect to vaccine education. We hypothesize that the intervention will increase knowledge about routine immunization among CHWs and patients, increase vaccine acceptance, intent-to-vaccinate, and vaccination rates among patients in the treatment group.

DETAILED DESCRIPTION:
Background:

Immunization programs in Sub-Saharan Africa have made progress in recent decades, yet coverage remains low overall for some childhood vaccines. Immunization is one of the most powerful and cost effective public health interventions. In addition to saving lives, vaccination can greatly reduce the burden of illness and disability from vaccine preventable diseases, and contribute to improving child health and welfare, as well as reducing hospitalization costs. Yet, globally, mistrust in childhood vaccinations increased during the COVID-19 pandemic. Vaccine hesitancy in Kenya is driven by multiple interrelated and interconnected factors, including mistrust in health systems and vaccine misinformation which has grown during the global COVID-19 pandemic.

Community Health Workers (CHWs) are vital to global vaccination efforts, both in the distribution and logistical support, but also in promoting vaccine acceptance. Now more than ever, CHWs face barriers as vaccine educators including the proliferation of misinformation, lack of reliable, up-to-date information, and limited training in effective communication.

Aim:

Researchers at Stanford University's Center for Health Education and the Lwala Community Health Alliance are partnering to investigate how to better support CHWs to improve routine vaccination rates in high-need areas by testing a two-part intervention. The first part of the intervention is a digital training provided to CHWs, which includes videos and job aids on vaccine education. The second part of the intervention is a patient-facing chatbot that is designed to provide patients with key information about routine immunizations with the intent of increasing patient knowledge about vaccines, vaccine acceptance, and vaccination rates.

Methods:

To test the effectiveness of training and equipping CHWs with the digital training and chatbot tool, study researchers will conduct a cluster randomized trial in the two focal subcounties in Migori County (Awendo and Nyatike) that the Lwala Community Health Alliance has identified as high need with respect to vaccine education. Lwala survey data suggest that between 20-25 percent of children under 5 years have not received routine immunizations in these two sub-counties. Early anecdotal data has shown that there are additional barriers and vaccine hesitancy concerns with the rollout of the new malaria vaccine.

CHWs in the focal subcounties are organized into regional administrative units known as Community Health Units (CHUs). Training is provided at regularly scheduled CHU meetings attended by CHWs on a regular basis. The research team will randomize CHUs (Awendo/ 31 CHUs and Nyatike/ 48 CHUs) into a treatment arm in which CHWs receive the training and chatbot tool and a control arm in which CHWs receive neither. The CHWs will be blinded to treatment assignment and informed that they are taking part in a study to understand the CHW experiences and their communication with patients. Randomization will be stratified by geographic units (wards) and whether a health facility is available in the ward.

The participants in the treatment group will receive the intervention at the start of the study, while the participants in the control group will receive upon conclusion of the study, which will allow for the comparison of knowledge, beliefs and vaccination rates with a group that is controlled for bias introduced by time. The duration of the study for participants will be roughly four months, which will allow CHWs ample time to introduce the chatbot to eligible patients and provide patients with time to use the chatbot to inform their vaccine decision making.

Intervention:

The intervention is being developed by the Stanford Center for Health Education Digital Medic Initiative in collaboration with Lwala Community Health Alliance. The first part of the intervention is a digital training provided to CHWs, which includes videos and job aids on vaccine education to support patient communication. The second part of the intervention is a patient-facing chatbot designed to provide key information about routine immunization that CHWs can share with their patients through the social media and messenger application, WhatsApp.

The Stanford team has led the production of the video content, job aids, and chatbot design. The Lwala team has partnered in intervention design and development at all stages including script writing, piloting, and checking for relevance and resonance of educational content. The video content addresses reasons to vaccinate, vaccine misperceptions, side effects, and other barriers to improve childhood vaccination uptake. The video content is complemented by a set of infographic job aids for CHWs to share with their patients to encourage childhood immunization uptake. Content will be available in English and Dholuo.

Data collection:

Treatment and control CHWs will complete a baseline and endline survey administered at the same time. The baseline survey will include demographic questions and questions about CHWs' work experience including their perceptions of vaccine safety and effectiveness and preparedness to educate patients about complex health topics including childhood immunization. The endline survey will include a knowledge assessment drawn from the training content, as well as measures of CHW vaccine acceptance and preparedness to educate patients about childhood immunization. A subsample of patients will be surveyed at endline from both the treatment and control groups. The patient survey will include demographic questions and questions about patients' knowledge and beliefs about childhood immunization, intent-to-vaccinate and vaccination status among household members.

Data Analysis:

The primary analysis will be based on intention-to-treat at the CHU unit. The analysis will include randomization strata fixed effects and control for baseline covariates to improve precision of estimates.

ELIGIBILITY:
Inclusion Criteria:

* CHWs identified by Lwala Community Health Alliance in study area
* Patients with children in the household of eligible age for routine immunization

Exclusion Criteria:

- Patients without children in the household of eligible age for routine immunization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 795 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
CHW vaccine knowledge | Collected after roughly 1 month of exposure to the training content
  Knowledge about routine childhood vaccines based on a set of 15 knowledge questions draw directly from the digital training
CHW vaccine beliefs | Collected after roughly 1 month of exposure to the training content
  Set of 5 Likert scale questions about beliefs about routine childhood vaccines regarding 1) the safety of childhood vaccines, 2) the effectiveness of childhood vaccines, 3) whether children should receive the new Malaria vaccine, 4) whether children receive too many vaccines, and 5) whether vaccination is compatible with one's personal beliefs.
CHW vaccine education preparedness | Collected after roughly 1 month of exposure to the training content
  Set of 5 Likert scale questions about preparedness to educate patients about routine childhood vaccines including 1) preparedness to answer patient questions, 2) preparedness to explain complex health topics including immunization to patients, 3) adequate access to information about vaccines and the diseases they prevent, 4) preparedness to explain the need for so many childhood vaccines, and 5) preparedness to alleviate patients' fears about vaccination.
Patient vaccine knowledge | Collected roughly 4-6 months from CHW first exposure to the training content
  Knowledge about routine childhood vaccines based on a set of 15 knowledge questions draw directly from the digital training
Patient vaccine beliefs | Collected roughly 4-6 months from CHW first exposure to the training content
  Set of 5 Likert scale questions about beliefs about routine childhood vaccines regarding 1) the safety of childhood vaccines, 2) the effectiveness of childhood vaccines, 3) whether children should receive the new Malaria vaccine, 4) whether children receive too many vaccines, and 5) whether vaccination is compatible with one's personal beliefs.
Patient vaccination uptake | Collected roughly 6 months from CHW first exposure to the training content
  Vaccination uptake among patients of treatment CHWs measured by CHW records, patient self reports, and administrative health records (where available)

SECONDARY OUTCOMES:
CHW perceptions of patient vaccine beliefs | Collected after roughly 1 month of exposure to the training content
  Set of 6 Likert scale questions posted to CHWs about the beliefs of their patients including whether their patients 1) believe vaccines are safe, 2) believe vaccines are important, 3) know when you bring children to clinic to receive vaccinations, 4) believe that all doses are important for children to receive, 5) are fearful of adverse vaccine side effects, and 6) are fearful of long-term impact of vaccines on their children.

CONTACTS AND LOCATIONS:
Locations (1):
- Lwala Community Health Alliance, Rongo, Kenya

IPD SHARING:
Plan to Share IPD: Undecided